CLINICAL TRIAL: NCT00540397
Title: Traditional Chinese Medicine Etiological Study on the Theory of XuSunShengJi in Liver Cirrhosis
Brief Title: TCM Etiological Study on the Theory of XuSunShengJi in Liver Cirrhosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai University of Traditional Chinese Medicine (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2006CB504801
Record Dates: First submitted 2007-10-05; First posted 2007-10-08 (Estimated); Last update posted 2007-10-08 (Estimated); Status verified 2007-10

CONDITIONS: Liver Cirrhosis
MeSH Terms: conditions — Liver Cirrhosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Fuzhenghuayu Tablet, Huangqi Decoction Granule

SUMMARY:
To Elucidate and Confirm the Theory of XuSunShengJi in the Traditional Chinese Medicine Etiological Pathogenesis of Liver Cirrhosis.

ELIGIBILITY:
Inclusion Criteria:

* With 6 month of chronic liver disease history, and positive serum HBsAg

Exclusion Criteria:

* Other chronic hepatitis and liver cirrhosis of non-hepatitis B

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Ping Liu, Professor, Principal Investigator — Shanghai University of Traditional Chinese Medicine
Locations (1):
- Shuguang Hospital Affiliated to Shanghai University of Traditional Chinese Medicine, Shanghai, Shanghai Municipality, China